CLINICAL TRIAL: NCT05089227
Title: Efficacy of Prolonged Anticoagulation for Primary Prevention of Venous Thromboembolic Disease in Autoimmune Hemolytic Anemia: a Prospective, Phase II, Randomized, Multicenter Study
Acronym: API-AHAI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Dijon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AUDIA PHRCI 2019
Record Dates: First submitted 2021-10-11; First posted 2021-10-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Prolonged Anticoagulation; Venous Thromboembolic Disease; Autoimmune Hemolytic Anemia
MeSH Terms: conditions — Anemia, Hemolytic, Autoimmune | interventions — Crisis Intervention

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- "intervention" group (Experimental)
  Interventions: Drug: treatment "intervention"; Biological: biological assessment
- "standard" group (Active Comparator)
  Interventions: Drug: treatment "standard"; Biological: biological assessment

INTERVENTIONS:
Drug: treatment "intervention" — for a total of 12 weeks, prophylactic heparin therapy during hospitalization followed by prophylactic oral anticoagulation with apixaban
  Arms: "intervention" group
Drug: treatment "standard" — during hospitalization prophylactic heparin therapy followed by management without prophylactic anticoagulation.
  Arms: "standard" group
Biological: biological assessment — CBC, reticulocytes, haptoglobin, LDH, bilirubin

SUMMARY:
Autoimmune hemolytic anemia (AIHA) is a rare autoimmune disease (incidence <1/100,000 population) responsible for the destruction of red blood cells by the host immune system, notably through the action of autoantibodies.

Apart from complications related to anemia, the occurrence of venous thromboembolism (VTE) in this population is frequent, estimated at 20-27%. The risk of VTE is highest during the period of hemolysis, especially during the first 3 months after the diagnosis of AIHA. This risk is 7.5 [4.7; 12.0] times greater than in the general population. No clinical predictive factor for VTE was identified and the usual factors (cancer, previous VTE, bed rest >3 days, surgery, age >70 years, heart or respiratory failure, myocardial infarction, stroke, obesity, hormone replacement therapy) were not considered. Several biological risk factors have been suggested (depth of anemia, bilirubin level, leukocyte count, antiphospholipid antibodies) but have not been confirmed in other studies.

AIHA is therefore a risk factor for VTE in its own right, and the National Diagnostic and Care Protocol (NDCP) recommends the implementation of VTE prevention during acute hemolysis (Grade C). However, the value of this prophylaxis has never been prospectively evaluated and its duration is empirical. In practice, low-molecular-weight heparin (LMWH) is generally used during "flare-ups" of AIHA (diagnosis and relapse) in hospitalized patients, but is rarely continued beyond the hospital phase when VTE also occurs in ambulatory patients.

Thus, we hypothesize that prolonged preventive anticoagulation during the 12-week risk period following diagnosis or relapse of AIHA could decrease the incidence of VTE.

In orthopedic surgery, this strategy has been proven to decrease VTE from 50% to 10-15%. In certain high-risk medical situations, prolonged prophylaxis with apixaban has been shown to decrease the occurrence of VTE from 10.2% to 4.2% in solid cancers4 and from 4-11% to 2% in myeloma.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged ≥ 18 years
* Patient with a diagnosis of primary or secondary autoimmune hemolytic anemia (AIHA) (infections, hematologic diseases, systemic diseases), according to the following criteria:
* Hemoglobin <12 g/dL
* and decreased haptoglobin (<0.4 g/L)
* and positive direct antiglobulin test (direct Coombs test) (IgG +/- C3d)
* Patient newly diagnosed or relapse
* Patient with an estimated life expectancy of more than 6 months
* Patient who provided free, written and informed consent

Exclusion Criteria:

* Patients with immediate symptomatic VTE, confirmed by appropriate complementary examinations (venous Doppler of the lower limbs, thoracic angioscanner or pulmonary scintigraphy).
* Patients on curative anticoagulation (venous thromboembolic disease, atrial fibrillation)
* Patient on dual antiaggregation treatment
* Patient with active bleeding
* Patient with a known condition or lesion at risk of bleeding
* Patient with ischemic stroke with hemorrhagic transformation within 6 months prior to inclusion
* Patient on preventive anticoagulation for 14 days or more
* Patient with a contraindication to apixaban:
* Known hypersensitivity to the molecule or to any of the excipients,,
* thrombocytopenia <100 G/L,
* kidney failure (glomerular filtration rate < 30 ml/min/1.73m²)
* Active liver disease (liver failure defined as Factor V <50% or INR >1.5, ALT elevation >2 times the upper limit of normal)
* Patients receiving concomitant CYP3A4 inducers (rifampin, phenytoin, carbamazepine, phenobarbital, St. John's Wort) or CYP3A4 inhibitors (azole antifungals, HIV protease inhibitors), if these therapies cannot be discontinued or modified
* Patients with a contraindication to enoxaparin:
* allergy to the drug
* history of heparin-induced thrombocytopenia
* Patient with cold agglutinin-related AHAI (C3d-positive ADT alone with identification of cold agglutinins)
* Patient with severe disorders of hemostasis:
* hypofibrinogenemia < 2 g/L,
* disseminated intravascular coagulation (APTT prolongation>1.2, and PT<50%, and thrombocytopenia<100 G/L, and D-Dimer >500 µg/L)
* hemophilia
* Patient whose clinical condition requires hospitalization in an intensive care unit
* Patient who has already participated in the study
* Patient not affiliated to national health insurance
* Patient under legal protection (curatorship, guardianship)
* Patient subject to a measure of legal protection
* Pregnant, parturient or breastfeeding women
* Patient with physiological capacity to procreate (having had her first menstrual period and not menopausal and not presenting permanent sterility (hysterectomy, bilateral salpingectomy, bilateral oophorectomy)) and unable to have effective contraception (i.e., provided by an estrogen-progestin oral contraceptive or progestogen, a contraceptive implant, an intrauterine device or a tubal ligation)
* Patient of legal age who is unable to provide consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-02-03 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Occurrence of clinical venous thromboembolic events (deep vein thrombosis (DVT) and pulmonary embolism (PE)) | 24 weeks after randomization
  defined by the presence of DVT confirmed by venous Doppler and/or PE confirmed by thoracic angioscan or ventilation/perfusion lung scintigraphy.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Dijon Bourgogne, Dijon, France